CLINICAL TRIAL: NCT00893451
Title: Does Vitamin D3 (Cholecalciferol) Supplementation Change Insulin Resistance in Patients With Chronic Kidney Disease?
Brief Title: Study of Vitamin D3 Supplementation in Patients With Chronic Kidney Disease
Acronym: VitaD-CKD1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Hamid Dezfoolian, MD, Dept. of kidney disease, Sahlgrenska University Hospital, Gothenburg, Sweden
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: VitaD-CKD1
Record Dates: First submitted 2009-05-05; First posted 2009-05-06 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2011-06

CONDITIONS: Chronic Kidney Disease; Insulin Resistance; Vitamin D Deficiency
Keywords: renal disease; renal impairment; chronic kidney disease stage 3-4; 25(OH) vitamin D; cholecalciferol; vitamin D deficiency; insulin resistance; insulin-glucose clamp; non-diabetic
MeSH Terms: conditions — Renal Insufficiency, Chronic; Insulin Resistance; Vitamin D Deficiency; Kidney Diseases; Renal Insufficiency | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): Vitamin D3 1600 IU orally twice daily
  Interventions: Drug: cholecalciferol (TillVal-D)
- B (Placebo Comparator): Placebo orally twice daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: cholecalciferol (TillVal-D) — In a randomized, two-way cross-over design participants will take vitamin D3 or placebo twice daily during treatment periods of 10 weeks separated by a washout period of 6 weeks.
  Other Names: TillVal-D, cholecalciferol, vitamin D3
  Arms: A
Drug: Placebo — Placebo orally twice daily
  Arms: B

SUMMARY:
The purpose of this study is to evaluate the impact of vitamin D3 supplementation on the insulin resistance in non-diabetic patients with chronic kidney disease (CKD) stages 3-4, vitamin D deficiency/insufficiency and elevated fasting serum insulin levels.

DETAILED DESCRIPTION:
Insulin resistance, i.e., reduction in insulin responsiveness with a decrease in glucose uptake in insulin target tissues (muscle and adipose tissue) is common in end-stage renal disease (ESRD), but is also present at earlier stages of renal disease with mild-moderate renal function impairment as well as in microalbuminuria and nephrotic syndrome.

Population-based cross-sectional studies have shown that low levels of vitamin D (25(OH) vitamin D) is associated with impaired glucose tolerance in subjects with normal renal function and that reduced renal function and 25(OH) vitamin D deficiency are independently associated with insulin resistance.

Vitamin D has well-known effects on calcium metabolism and skeletal mineralisation but recent experimental studies suggest that vitamin D in addition reduces several inflammatory mediators that are of importance in the development and progression of renal disease which also associated with insulin resistance such as TNF-α and IL-6.

This is a prospective, single-blind, explorative, randomized, placebo-controlled, single-centre, two-way cross-over study with two treatment periods of 10 weeks separated by a washout period of 6 weeks. Non-diabetic patients with chronic kidney disease (CKD) stage 3 and 4 (GFR 15-60 ml/min/1.73m2) who have low serum 25-OH-vitamin D levels (< 30 ng/mL) and elevated fasting serum insulin levels (>10 IU/L) will be randomized to receive either vitamin D3 (cholecalciferol) 3200U orally (tablets) daily or placebo.

Approximately 24 patients are going to complete the study. A pre-entry wash-out period of 6 weeks is needed for patents already on vitamin D treatment. An in vivo assessment of insulin secretion and insulin sensitivity will be made by insulin-glucose clamp at the end of each treatment period.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age older than 18 years
2. Non-diabetic chronic kidney disease stage 3 and 4 (GFR 15-60 ml/min/1.73 m2)
3. Serum 25(OH) vitamin D < 30 ng/mL (75 nmol/L)
4. Fasting S-insulin > 30 IU/L
5. Written informed consent before entered into study

Exclusion Criteria:

1. Patients with current significant, major or unstable cardio-cerebrovascular, infection, respiratory, gastrointestinal or other major disease and risks according to the judgment made by the investigator
2. Patients with type 1 or type 2 Diabetes
3. Current severe thyrotoxicosis or other endocrine disease
4. Granulomatous disease, such as sarcoidosis and tuberculosis
5. Patients who are intended to receive hemodialysis (HD), peritoneal dialysis (PD) or being kidney transplanted during the course of study (9 months)
6. Concomitant use of corticosteroids (except for inhalation or topical use) or other immunosuppressive medication
7. Treatment with biphosphonate during last two years
8. S-Calcium > 2.70 mmol/L (0.68 mg/dl)
9. PTH intact < 75 ng/L (8.25 nmol/L) or > 800 ng/L (88 nmol/L)
10. Proteinuria > 3.5 g/24 hours
11. Alcohol or drug abuse or any condition associated with poor compliance
12. Blood donors
13. Women of childbearing potential, desired pregnancy, pregnancy or lactation within the study period
14. Allergy or intolerance to cholecalciferol supplementation (TillVal D®) or other constituents
15. Participation in a clinical trial evaluating an investigational drug in the last 12 weeks prior to inclusion to this trial
16. History of kidney stones
17. History of chronic hepatitis or liver enzymes (ASAT or ALAT) more than 2.5 times the upper limit of normal
18. Gastrointestinal disease resulting in significant gastrointestinal dysfunction or malabsorption
19. Use of medications known to interact with vitamin D metabolism such as cholestyramine, phenytoin, digitalis and antacids
20. Planned vacation with "high sun exposure" during the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2009-09; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Change in M-value (mg/kg lean body mass/min) assessed by insulin-glucose clamp | at week 26

SECONDARY OUTCOMES:
Change in systolic- and diastolic blood pressure | at week 26
Change in PTH secretion and its fragments assessed by PTH, CAP-PTH, CIP-PTH | at week 26
Change in insulin secretion assessed by intravenous glucose tolerance test | at week 26
Change in urinary excretion of albumin (UAE) assessed by 24 hour collection | at week 26

CONTACTS AND LOCATIONS:
Overall Officials: Hamid R Dezfoolian, MD, Principal Investigator — Sahlgrenska University Hospital
Locations (1):
- Department of Kidney diseases, Sahlgrenska University Hospital, Gothenburg, Sweden